CLINICAL TRIAL: NCT02744404
Title: Evaluation of the Clinical Impact of Point-of-Care HIV Early Infant Diagnostic Technologies
Brief Title: Point of Care Early Infant Diagnosis Patient Impact Study
Status: Completed | Type: Observational
Sponsor: Clinton Health Access Initiative Inc. (Other)
Collaborators: Ministry of Health, Malawi (Other Government); UNICEF (Other)
Responsible Party: Sponsor
Other Study IDs: Malawi POC EID
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- POC EID: Point of Care Early Infant Diagnosis qualitative technologies (Alere q) will be implemented. Sample collection and testing will happen in the same location within the health care facility.
  Interventions: Device: POC EID
- Laboratory-based testing: Conventional laboratory-based testing using the Abbott m2000 technology will continue to be used per standard of care in Malawi. Dried blood spot samples will be collected at health care facilities and transported within the national network to centralized laboratories for testing.

INTERVENTIONS:
Device: POC EID
  Groups: POC EID

SUMMARY:
In Malawi, early infant HIV diagnosis (EID, i.e. HIV screening of infants under 18 months of age) is conducted using molecular diagnostics at central laboratories. However, test volumes are growing and many parts of the country do not have close or easy access to laboratories. Test samples are transported over large distances and this can introduce testing delays, especially for patients in rural and remote areas of the country. There are growing numbers of high quality Point-Of-Care (POC) diagnostic technologies available and there is increasing interest in using these technologies to alleviate critical testing needs. This protocol describes an observational study looking at the patient impact of implementing POC EID technologies within the routine standard of care at seven facilities.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 12 months of age
* Clinical or other indication for an EID test (screen or confirmation), such as birth to an HIV-positive mother

Exclusion Criteria:

* Older than 12 months of age
* Serious medical conditions which would make testing dangerous for the infant, or disrupt the accuracy of normal laboratory analysis and its interpretation
* Already initiated ART

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will be mother-infant pairs from the general population attending the seven clinics for routine HIV-related, PMTCT and post-natal care services. Study subjects will be infants from mother-infant pairs presenting consecutively to the clinic for EID testing per the national EID guidelines during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1752 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
ART initiation retention | 6-9 months
  Proportion of HIV-positive infants initiated on anti-retroviral therapy

SECONDARY OUTCOMES:
Test turnaround time | 6-9 months
  Number of days from testing to result being received by the health care facility
Tests received | 6-9 months
  Proportion of tests received by the health care facility

CONTACTS AND LOCATIONS:
Locations (7):
- Malawi (7):
  - Kamuzu Central Hospital, Lilongwe
  - Machinga District Hospital, Liwonde
  - Mzuzu Central Hospital, Mzuzu
  - Nsanama Health Center, Nsanama
  - Ntaja Health Center, Ntaja
  - Ntcheu District Hospital, Ntcheu
  - Migowi Health Center, Phalombe